CLINICAL TRIAL: NCT06017973
Title: The Role of Cerebral Functional, Structural and Spectral Imaging in the Diagnosis, Management and Prognosis of Status Epilepticus: a Prospective Study in Patients with the Ictal-interictal Continuum
Brief Title: The Role of Imaging in the Diagnosis, Management and Prognosis of Possible Non-convulsive Status Epilepticus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S67933
Record Dates: First submitted 2023-07-11; First posted 2023-08-30 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Status Epilepticus; Ictal-interictal Continuum; Positron-emission Tomography; Perfusion Weighted MRI; Perfusion CT
Keywords: possible non-convulsive status epilepticus; ictal-interictal continuum; EEG; MRI; FDG-PET; CT perfusion
MeSH Terms: conditions — Status Epilepticus | interventions — Cerebrovascular Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Possible non-convulsive status epilepticus with ictal-interictal continuum EEG patterns (Other): Patients with a possible non-convulsive status epilepticus, according to American Clinical Neurophysiology Criteria (ACNS) (2021).
  Interventions: Diagnostic Test: MRI scan including arterial spin labelling of the brain; Diagnostic Test: CT perfusion scan of the brain; Diagnostic Test: FDG-PET scan of the brain
- Healthy control subjects (Other): Healthy control subjects.
  Interventions: Diagnostic Test: MRI scan including arterial spin labelling of the brain; Diagnostic Test: CT perfusion scan of the brain; Diagnostic Test: FDG-PET scan of the brain

INTERVENTIONS:
Diagnostic Test: MRI scan including arterial spin labelling of the brain — Arterial Spin Labelling sequence, T2-weighted FLAIR images and T1-weighted images and diffusion weighted imaging sequence will be recorded
  Other Names: Brain perfusion
Diagnostic Test: CT perfusion scan of the brain — Siemens Naeotom Alpha with quantum technology (photon-counting)
  Other Names: Brain perfusion
Diagnostic Test: FDG-PET scan of the brain — An FDG-PET scan will be acquired on a GE Signa 3T PET-MR scanner. FDG-PET images will be assessed for focal hypermetabolism, including semiquantitative analysis of the maximal standard uptake value (SUVmax) relative to the SUVmax of the pons (SUVr pons)
  Other Names: Brain metabolism

SUMMARY:
The investigators propose a prospective study of 20 control subjects and 180 consecutive patients with possible non-convulsive status epilepticus (NCSE). The investigators will obtain three functional images of the brain:

1. Fluorodeoxyglucose positron emission tomography (FDG-PET)
2. Perfusion (and structural) magnetic resonance (MR) images
3. Computed tomography (CT) perfusion.

Brain hypermetabolism/hyperperfusion is a strong argument to confirm a diagnosis of non-convulsive status epilepticus.

The aim is to determine which of the three functional imaging techniques is the most sensitive and easy to obtain in the detection of hypermetabolism/hyperperfusion. The investigators will determine which EEG patterns are associated with hypermetabolism/perfusion.

The investigators will further study and describe the management with antiseizure medication and outcome of the group with possible non-convulsive status epilepticus WITH hypermetabolism/hyperperfusion versus the group with possible non-convulsive status epilpticus WITHOUT hypermetabolism/hyperperfusion.

The investigators will make recommendations for an imaging protocol in possible NCSE for widespread use. The aim is to offer guidelines to incorporate imaging in the diagnosis, management and prognosis of NCSE in patients with the ictal-interictal continuum.

ELIGIBILITY:
Inclusion Criteria:

- The patient has possible non-convulsive status epilepticus with scalp or invasive EEG with ictal-interictal continuum patterns on EEG

Exclusion Criteria:

* The patient has a contra-indication for MRI such as metal implants
* The patient has contrast sensitivity
* The patiensuffers from claustrophobia or cannot tolerate confinement during PET-MRI scanning procedures

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of MRI arterial spin labelling, CT perfusion and FDG-PET of the brain to detect hyperperfusion/hypermetabolism in possible non-convulsive status epilepticus | Day 1
  The investigators will determine which diagnostic test (MRI, CT or FDG-PET) is most sensitive in detecting hyperperfusion/hypermetabolism in possible non-convulsive status epilepticus to confirm a diagnosis of non-convulsive status epilepticus
Correlation between FREQUENCY of ictal-interictal EEG patterns within 30 minutes after FDG-PET injection and standardised uptake value on FDG-PET. | Day 1
  The investigators will assess the correlation between standardised uptake value of the cerebral hypermetabolic region and the frequency of ictal-interictal EEG patterns within 30 minutes after injection of FDG. The frequency of ictal-interictal EEG patterns will be scored semi-quantitatively based on the American Clinical Neurophysiology Criteria (ACNS) criteria (2021).
Correlation between PREVALENCE of ictal-interictal EEG patterns on EEG within 30 minutes after FDG-PET injection and standardised uptake value on FDG-PET. | Day 1
  The investigators will assess the correlation between standardised uptake value of the cerebral hypermetabolic region and the prevalence of ictal-interictal EEG patterns within 30 minutes after injection of FDG. The prevalence of ictal-interictal EEG patterns will be scored semi-quantitatively based on the American Clinical Neurophysiology Criteria (ACNS) (2021)
The seizure freedom of patients with hypermetabolism compared to those with hypometabolism within 24 hours after undergoing an FDG-PET scan. | Day 1
  The investigators will assess the seizure freedom of patients in the hypermetabolic vs hypometabolic group. Patients will receive video EEG-monitoring for 24 hours after FDG-PET. Seizures will be defined according to current American Clinical Neurophysiology Criteria (ACNS) (2021) based on electrographic and clinical data. Hypermetabolism/hypometabolism will be qualitatively scored by a trained nuclearist.

SECONDARY OUTCOMES:
Correlation between SHARPNESS of ictal-interictal EEG patterns on EEG within 30 minutes after FDG-PET injection and standardised uptake value on FDG-PET. | Day 1
  The investigators will assess the correlation between standardised uptake value of the cerebral hypermetabolic region and the sharpness of ictal-interictal EEG patterns within 30 minutes after injection of FDG. The sharpness of ictal-interictal EEG patterns will be scored semi-quantitatively based on the American Clinical Neurophysiology Criteria (ACNS) (2021)
Correlation between AMPLITUDE of ictal-interictal EEG patterns within 30 minutes after FDG-PET injection and standardised uptake value on FDG-PET | Day 1
  The investigators will assess the correlation between standardised uptake value of the cerebral hypermetabolic region and the amplitude of ictal-interictal EEG patterns within 30 minutes after injection of FDG. The amplitude of ictal-interictal EEG patterns will be scored semi-quantitatively based on the American Clinical Neurophysiology Criteria (ACNS) (2021)
Correlation between EVOLUTION of ictal-interictal EEG patterns on EEG within 30 minutes after FDG-PET injection and standardised uptake value on FDG-PET. | Day 1
  The investigators will assess the correlation between standardised uptake value of the cerebral hypermetabolic region and evolution of ictal-interictal EEG patterns within 30 minutes after injection of FDG (i.e. static, fluctuating or evolving). The presence of fluctuation and evolution of ictal-interictal EEG patterns will be scored based on the American Clinical Neurophysiology Criteria (ACNS) (2021)
Functional imaging in possible non-convulsive status epilepticus and INTERICTAL BURDEN | Day 7
  The investigators will compare interictal burden, defined as a percentage of ictal-interictal EEG patterns during continuous EEG monitoring, in the group with possible non-convulsive status epilepticus WITH hypermetabolism/hyperperfusion versus the group with possible non-convulsive status epilepticus WITHOUT hypermetabolism/hyperperfusion
Functional imaging in possible non-convulsive status epilepticus and ANTISEIZURE MEDICATION (ASM) | Day 30
  The investigators will document all changes in antiseizure medication and compare these in the group with possible non-convulsive status epilepticus WITH hypermetabolism/hyperperfusion versus the group with possible non-convulsive status epilepticus WITHOUT hypermetabolism/hyperperfusion
Functional imaging in possible non-convulsive status epilepticus and OUTCOME | Day 7
  The investigators will compare modified rankin scale (mRS) (0: no symptoms, 1: no significant disability, 2: slight disability, 3: moderate disability, 4: moderately severe disability, 5: severe disability and 6: death) at 7 days in the group with possible non-convulsive status epilepticus WITH hypermetabolism/hyperperfusion versus the group with possible non-convulsive status epilepticus WITHOUT hypermetabolism/hyperperfusion
Functional imaging in possible non-convulsive status epilepticus and OUTCOME | Day 30
  The investigators will compare modified rankin scale (mRS) (0: no symptoms, 1: no significant disability, 2: slight disability, 3: moderate disability, 4: moderately severe disability, 5: severe disability and 6: death) at 30 days in the group with possible non-convulsive status epilepticus WITH hypermetabolism/hyperperfusion versus the group with possible non-convulsive status epilepticus WITHOUT hypermetabolism/hyperperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Paesschen, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, department of Neurology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Our original imaging and annotated EEG data will be made available to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be made available after publication of our results. There is no end date.
Access Criteria: Proposals should be directed to Jeroen.gijs@uzleuven.be. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Trinka E, Cock H, Hesdorffer D, Rossetti AO, Scheffer IE, Shinnar S, Shorvon S, Lowenstein DH. A definition and classification of status epilepticus--Report of the ILAE Task Force on Classification of Status Epilepticus. Epilepsia. 2015 Oct;56(10):1515-23. doi: 10.1111/epi.13121. Epub 2015 Sep 4. PMID 26336950
- [Background] Hirsch LJ, Fong MWK, Leitinger M, LaRoche SM, Beniczky S, Abend NS, Lee JW, Wusthoff CJ, Hahn CD, Westover MB, Gerard EE, Herman ST, Haider HA, Osman G, Rodriguez-Ruiz A, Maciel CB, Gilmore EJ, Fernandez A, Rosenthal ES, Claassen J, Husain AM, Yoo JY, So EL, Kaplan PW, Nuwer MR, van Putten M, Sutter R, Drislane FW, Trinka E, Gaspard N. American Clinical Neurophysiology Society's Standardized Critical Care EEG Terminology: 2021 Version. J Clin Neurophysiol. 2021 Jan 1;38(1):1-29. doi: 10.1097/WNP.0000000000000806. No abstract available. PMID 33475321
- [Background] Cormier J, Maciel CB, Gilmore EJ. Ictal-Interictal Continuum: When to Worry About the Continuous Electroencephalography Pattern. Semin Respir Crit Care Med. 2017 Dec;38(6):793-806. doi: 10.1055/s-0037-1607987. Epub 2017 Dec 20. PMID 29262437
- [Background] Rubinos C, Reynolds AS, Claassen J. The Ictal-Interictal Continuum: To Treat or Not to Treat (and How)? Neurocrit Care. 2018 Aug;29(1):3-8. doi: 10.1007/s12028-017-0477-5. PMID 29139014
- [Background] Osman GM, Araujo DF, Maciel CB. Ictal Interictal Continuum Patterns. Curr Treat Options Neurol. 2018 Apr 18;20(5):15. doi: 10.1007/s11940-018-0500-y. PMID 29666958
- [Background] Rodriguez Ruiz A, Vlachy J, Lee JW, Gilmore EJ, Ayer T, Haider HA, Gaspard N, Ehrenberg JA, Tolchin B, Fantaneanu TA, Fernandez A, Hirsch LJ, LaRoche S; Critical Care EEG Monitoring Research Consortium. Association of Periodic and Rhythmic Electroencephalographic Patterns With Seizures in Critically Ill Patients. JAMA Neurol. 2017 Feb 1;74(2):181-188. doi: 10.1001/jamaneurol.2016.4990. PMID 27992625
- [Background] Struck AF, Westover MB, Hall LT, Deck GM, Cole AJ, Rosenthal ES. Metabolic Correlates of the Ictal-Interictal Continuum: FDG-PET During Continuous EEG. Neurocrit Care. 2016 Jun;24(3):324-31. doi: 10.1007/s12028-016-0245-y. PMID 27169855
- [Background] Subramaniam T, Jain A, Hall LT, Cole AJ, Westover MB, Rosenthal ES, Struck AF. Lateralized periodic discharges frequency correlates with glucose metabolism. Neurology. 2019 Feb 12;92(7):e670-e674. doi: 10.1212/WNL.0000000000006903. Epub 2019 Jan 11. PMID 30635488
- [Background] Venkatraman A, Khawaja A, Bag AK, Mirza M, Szaflarski JP, Pati SBB. Perfusion MRI Can Impact Treatment Decision in Ictal-Interictal Continuum. J Clin Neurophysiol. 2017 Jul;34(4):e15-e18. doi: 10.1097/WNP.0000000000000350. PMID 27749504
- [Background] Gugger JJ, Llinas RH, Kaplan PW. The role of CT perfusion in the evaluation of seizures, the post-ictal state, and status epilepticus. Epilepsy Res. 2020 Jan;159:106256. doi: 10.1016/j.eplepsyres.2019.106256. Epub 2019 Dec 12. PMID 31862478
- [Background] Trinka E, Leitinger M. Management of Status Epilepticus, Refractory Status Epilepticus, and Super-refractory Status Epilepticus. Continuum (Minneap Minn). 2022 Apr 1;28(2):559-602. doi: 10.1212/CON.0000000000001103. PMID 35393970